CLINICAL TRIAL: NCT03712150
Title: Role of Genetic Polymorphism in Neuroplasticity Involved in Dysphagia Recovery- Part 2
Brief Title: Effects of Gene Polymorphism After Transcranial Cranial Direct Current Stimulation on the Corticobulbar Excitability
Status: Completed | Type: Observational
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Sun Im, Sun Im, Assistant Professor, The Catholic University of Korea, The Catholic University of Korea
Other Study IDs: HC18TNSV0061
Record Dates: First submitted 2018-10-10; First posted 2018-10-19 (Actual); Last update posted 2019-11-07 (Actual); Status verified 2019-11

CONDITIONS: Healthy
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — DNA of gene polymorphism from the Polymorphisms in brain-derived neurotrophic factor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy: Healthy adults
  - Participants will receive single session of tdcs after application
  Interventions: Device: tdcs

INTERVENTIONS:
Device: tdcs — application of optimised parameters of tDCS (anodal stimulation, 1.5 mA, 10 min) over the unconditioned hemisphere reverses the brain and behavioural consequences of inhibitory pre-conditioning

SUMMARY:
This study aims to examine the effects of transcranial direct current stimulation at corticobulbar excitability in individuals with different gene polymorphism.

DETAILED DESCRIPTION:
The effects of TDCS on corticobulbar excitability of the brain after inhibitory pre-conditioning will be compared in patients with different BDNF phenotypes

ELIGIBILITY:
Inclusion Criteria:

* Age 19-40 years
* Informed consent

Exclusion Criteria:

* History of epilepsy
* Presence of cardiac pacemaker
* previous brain surgery
* previous swallowing problems
* current use of medication which acts on the central nervous system
* presence of implanted metal intracranially

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy young volunteers
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-11-10 (Actual); Primary Completion 2019-06-08 (Actual); Study Completion 2019-08-08 (Actual)

PRIMARY OUTCOMES:
Brain corticobulbar excitability | Immediately after single conditioning the brain
  Change of Brain corticobulbar excitability by motor evoked potentials

SECONDARY OUTCOMES:
Tongue pressure measurement- | Immediate after single conditioning the brain
  Change of tongue pressure measurement by Intra oral pressure assessment
Electrophysiological responses of swallowing - | Immediate after single conditioning the brain
  Change of Electrophysiological responses of swallowing - With the use of a laryngeal transducer, will measure the mylohyoid amplitude

CONTACTS AND LOCATIONS:
Overall Officials: Sun Im, MD PhD, Principal Investigator — The Catholic University of Korea
Locations (2):
- South Korea (2):
  - Department of Rehabilitation Medicine, Bucheon-si, Bucheonshi
  - Department of Rehabilitation Medicine Bucheon St Mary's Hospital, Catholic University of Korea, College of Medicine, Bucheon-si, Kyounggido

IPD SHARING:
Plan to Share IPD: No